CLINICAL TRIAL: NCT00121134
Title: Anti-Angiogenesis Treatment After Preoperative Chemotherapy: A Pilot Study in Women With Operable Breast Cancer
Brief Title: Bevacizumab With or Without Cyclophosphamide and Methotrexate: A Pilot Study in Women With Operable Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harold J. Burstein, MD, PhD (Other)
Collaborators: Genentech, Inc. (Industry); Beth Israel Deaconess Medical Center (Other); Indiana University School of Medicine (Other); University of California, San Francisco (Other); University of North Carolina (Other)
Responsible Party: Sponsor-Investigator, Harold J. Burstein, MD, PhD, Associate Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-055
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: Bevacizumab; Metronomic Chemotherapy; Breast Cancer Stages II-III; Invasive breast cancer stages II-III
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Cyclophosphamide; Methotrexate; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): Bevacizumab Alone
  Interventions: Drug: Bevacizumab
- Group B (Experimental): Bevacizumab with cyclophosphamide and methotrexate
  Interventions: Drug: Bevacizumab; Drug: Cyclophosphamide; Drug: Methotrexate
- Group C (Experimental): capecitabine, 14 days on/7 days off scheduling, and bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Capecitabine
- Group D (Experimental): capecitabine 7 days on/7 days off scheduling, and bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab — Group A: Once every 3 weeks for 12 months Group B: Once every 3 weeks for 12 months
  Other Names: Avastin
Drug: Cyclophosphamide — Once a day for 6 months
  Other Names: Cytoxan
  Arms: Group B
Drug: Methotrexate — Twice daily for the first two days of every week for 6 months
  Other Names: amethopterin
  Arms: Group B
Drug: Capecitabine — Capecitabine: 2000 mg/m2 a day, on Days 1-14 of a 21 day cycle, for at total of 6 cycles (18 weeks)
  Bevacizumab: 15 mg/kg IV day 1 every 3 weeks x 1 year (17 cycles)
  Other Names: Xeloda
  Arms: Group C; Group D

SUMMARY:
The purpose of this research study is to study the effects (good and bad) of bevacizumab alone, bevacizumab with low-dose continuous chemotherapy (called metronomic chemotherapy), or bevacizumab with capecitabine, on you and your cancer. The goals of the study will be to:

* Examine the safety of these drugs
* See how easy or difficult it is to be treated with them
* Monitor for any signs of recurrent cancer
* Look at blood markers that might indicate how the treatment is working

DETAILED DESCRIPTION:
This study is broken into 4 groups (A, B, C, and D). Enrollment closed to all groups in May 2008.

The first forty subjects (Group A) in this study were treated with Bevacizumab only, which is given through a vein over 1-2 hours every 3 weeks, for a total of approximately 12 months (17 cycles). Each cycle consists of 3 weeks.

The next forty subjects (Group B) were treated with Bevacizumab and metronomic CM chemotherapy. These subjects took cyclophosphamide (1 pill by mouth every day), methotrexate, (1 pill taken by mouth twice a day for the first two days of each week) and Bevacizumab (once every 3 weeks). The treatments with cyclophosphamide, methotrexate and Bevacizumab will continue for approximately 6 months (8 cycles). Then for the next 6 months, they received Bevacizumab treatments only. The total time on this study will be about 12 months (17 cycles).

The next forty subjects (Group C) were treated with Bevacizumab and Capecitabine chemotherapy. These subjects took Capecitabine pills twice a day for 14 days, then one week of rest, to complete a 21-day cycle. There will be a total of 6 cycles of Capecitabine, meaning 18 weeks of treatment with both Capecitabine and Bevacizumab. Then received Bevacizumab treatments only (11 cycles) to complete 12 months of therapy. Total duration of your treatment will be about 12 months or 17 cycles of therapy.

The last forty subjects (Group D) are being treated with Bevacizumab and Capecitabine chemotherapy on a different schedule. These subjects will take Capecitabine pills twice a day for 7 days, then one week of rest and repeat this for a total of 24 weeks (6 cycles). Each cycle will last for 4 weeks (28 days). There will be a total of 6 cycles of Capecitabine, meaning 24 weeks of treatment with both Capecitabine and Bevacizumab. Bevacizumab will be given every two weeks for a total of 24 weeks (6 cycles). Then they will receive Bevacizumab treatments only, every 3 weeks for additional 27 weeks (9 cycles) to complete 12 months of therapy. For the last 9 cycles of Bevacizumab therapy each cycle will consist of 3 weeks. Total duration of treatment will be about 12 months or 15 cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, preoperative stages II-III per AJCC 6th edition, based on baseline evaluation by clinical examination and/or breast imaging
* Patients must have completed preoperative (neoadjuvant) chemotherapy with a standard chemotherapy regimen. No more chemotherapy should be planned.
* Patients must have completed definitive resection of primary tumor with adequate excision of gross disease.
* For patients receiving adjuvant radiation therapy, treatment must be completed prior to initiation of protocol therapy.
* Patients must have the presence of significant residual invasive disease on pathologic review following their preoperative chemotherapy.
* LVEF > institutional limits of normal after preoperative chemotherapy, as assessed by ECHO or nuclear medicine gated study, within 30 days prior to initiating protocol-based treatment.
* ECOG performance status 0-1

Exclusion Criteria:

* Inadequate organ function, as measured by laboratory assessment after preoperative chemotherapy and within 14 days of beginning protocol-based treatment
* Patients with metastatic disease are ineligible.
* Known HIV infection
* Patients may not be pregnant, expect to become pregnant, plan to conceive a child while on study, or breastfeeding
* Uncontrolled intercurrent illness
* Non-healing wounds or major surgical procedures (such as breast surgery) other than that for venous access device or diagnostic study are not permitted within 28 day prior to enrollment
* History of abdominal fistula, GI perforation, intra-abdominal abscess, or serious, non-healing wound, ulcer, or bone fracture within 6 months prior to initiating bevacizumab
* Patients with any history of arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular event (CVA), unstable angina, or myocardial infarction (MI) within the past 6 months. Patients with clinically significant peripheral arterial disease should also be excluded
* History of bleeding diathesis or coagulopathy
* History of grade 3 or 4 allergic reactions to compounds of similar chemical or biologic composition to cyclophosphamide (such as other alkylating agents) or methotrexate (such as other antimetabolites)
* Prior history of malignancy treated without curative intent, excluding nonmelanomatous skin cancer
* Patients with large or rapidly accumulating pleural or abdominal effusions
* Current use of anticoagulants is allowed as long as patients have been on a stable dose for more than two weeks with stable INR
* Chronic therapy with full dose aspirin (< 325 mg/day) or standard non-steroidal anti-inflammatory agents is allowed
* Patients may not receive other investigational agents while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2005-06; Primary Completion 2009-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold J Burstein, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of North Carolina, Durham, North Carolina

REFERENCES:
- [Derived] Trapani D, Jin Q, Miller KD, Rugo HS, Reeder-Hayes KE, Traina T, Abdou Y, Falkson C, Abramson V, Ligibel J, Chen W, Come S, Nohria A, Ryabin N, Tayob N, Tolaney SM, Burstein HJ, Mayer EL. Optimizing Postneoadjuvant Treatment of Residual Breast Cancer With Adjuvant Bevacizumab Alone, With Metronomic or Standard-Dose Chemotherapy: A Combined Analysis of DFCI 05-055 and DFCI 09-134/TBCRC 012/ABCDE Clinical Trials. Clin Breast Cancer. 2025 Jun;25(4):e419-e430.e5. doi: 10.1016/j.clbc.2024.12.018. Epub 2024 Dec 31. PMID 39890560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This sequential cohort phase II study was performed in the outpatient setting at four institutions between 2005 and 2008.
Pre-assignment Details: A total of 164 participants were registered to enroll in the trial , but only 162 participants initiated treatment. So the evaluable population is 162 participants.
Groups:
- Group A- Bevacizumab Alone: Bevacizumab 15 mg/kg every 3 wks for 1 year
- Group B-Bevacizumab+Cyclophosphamide+Methotrexate: Bevacizumab 15 mg/kg every 3 weeks for 1 year +Cyclophosphamide 50 mg orally daily for 6 months +methotrexate 2.5mg orally on day 1-2 each week for 6 months.
- Group C-Bevacizumab + Capcitabine(18 Wks): capecitabine 2000 mg/m2/day 14 days on/7 days off for 18 weeks, and bevacizumab 15 mg/kg every 3 weeks for 1 year
- Group D-bevacizumab + Capecitibine (24wks): capecitabine 2000 mg orally twice per day for 7 days on/7 days off for 24 weeks, and bevacizumab 15 mg/kg every 3 weeks for 1 year.
Period: Overall Study
Arm/Group | Group A- Bevacizumab Alone | Group B-Bevacizumab+Cyclophosphamide+Methotrexate | Group C-Bevacizumab + Capcitabine(18 Wks) | Group D-bevacizumab + Capecitibine (24wks)
Started | 40 | 41 | 41 | 40
Completed | 24 | 26 | 20 | 31
Not Completed | 16 | 15 | 21 | 9
Not completed — Progression of Disease | 5 | 3 | 4 | 2
Not completed — Toxicity | 4 | 7 | 13 | 5
Not completed — Physician Decision | 6 | 4 | 4 | 1
Not completed — Treatment Delay | 1 | 0 | 0 | 0
Not completed — Intercurrent Illness | 0 | 0 | 0 | 1
Not completed — Patient Personal Reasons | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A- Bevacizumab Alone | Group B-Bevacizumab+Cyclophosphamide+Methotrexate | Group C-Bevacizumab + Capcitabine(18 Wks) | Group D-bevacizumab + Capecitibine (24wks) | Total
Number analyzed (Participants) | 40 | 41 | 41 | 40 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.05 (10.04) | 48.83 (10.34) | 48.71 (10.34) | 49.55 (9.09) | 49.03 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 41 | 40 | 162
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 41 | 40 | 162

OUTCOME MEASURES:

1. Primary Outcome: The Completion Rate of 1 Year of Bevacizumab Therapy for All Four Cohorts
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Group A- Bevacizumab Alone | Group B-Bevacizumab+Cyclophosphamide+Methotrexate | Group C-Bevacizumab + Capcitabine(18 Wks) | Group D-bevacizumab + Capecitibine (24wks)
Number analyzed (Participants) | 40 | 41 | 41 | 40
percentage of participants | 60 | 58 | 49 | 76

ADVERSE EVENTS:
Arm/Group | Group A- Bevacizumab Alone | Group B-Bevacizumab+Cyclophosphamide+Methotrexate | Group C-Bevacizumab + Capcitabine(18 Wks) | Group D-bevacizumab + Capecitibine (24wks)
Serious Adverse Events (participants affected / at risk) | 1/40 | 3/41 | 1/41 | 1/40
Other Adverse Events (participants affected / at risk) | 40/40 | 41/41 | 41/41 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A- Bevacizumab Alone (N=40) | Group B-Bevacizumab+Cyclophosphamide+Methotrexate (N=41) | Group C-Bevacizumab + Capcitabine(18 Wks) (N=41) | Group D-bevacizumab + Capecitibine (24wks) (N=40)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lower GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A- Bevacizumab Alone (N=40) | Group B-Bevacizumab+Cyclophosphamide+Methotrexate (N=41) | Group C-Bevacizumab + Capcitabine(18 Wks) (N=41) | Group D-bevacizumab + Capecitibine (24wks) (N=40)
ALT, SGPT (Hepatobiliary disorders) | 3 (6) | 7 (8) | 2 (2) | 3 (7)
AST, SGOT (Hepatobiliary disorders) | 8 (17) | 12 (42) | 7 (12) | 3 (9)
Abdomen, pain (Gastrointestinal disorders) | 8 (10) | 2 (3) | 6 (15) | 1 (1)
Alkaline phosphatase (Hepatobiliary disorders) | 3 (12) | 2 (10) | 2 (2) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (17) | 0 (0) | 2 (2) | 3 (4)
Agitation (Psychiatric disorders) | 0 (0) | 1 (4) | 0 (0) | 2 (2)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (9) | 3 (6) | 2 (5)
Anorexia (Gastrointestinal disorders) | 6 (12) | 4 (12) | 8 (14) | 5 (15)
Anxiety (Psychiatric disorders) | 10 (33) | 8 (20) | 8 (34) | 7 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (7) | 0 (0) | 4 (9)
back,pain (Musculoskeletal and connective tissue disorders) | 9 (16) | 11 (31) | 9 (34) | 6 (13)
bicarbonate (Metabolism and nutrition disorders) | 0 (0) | 4 (11) | 1 (1) | 1 (1)
bilirubin (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (3) | 1 (2)
bone, pain (Musculoskeletal and connective tissue disorders) | 3 (7) | 2 (3) | 3 (12) | 2 (2)
breast,pain (Musculoskeletal and connective tissue disorders) | 6 (12) | 3 (22) | 3 (14) | 1 (1)
bruising (Blood and lymphatic system disorders) | 6 (12) | 3 (4) | 3 (11) | 1 (2)
buttock, pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Chelitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
chest wall, pain (Musculoskeletal and connective tissue disorders) | 4 (13) | 2 (6) | 1 (1) | 1 (1)
Chest/thoracic pain NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5) | 2 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 10 (25) | 5 (17) | 12 (31) | 13 (55)
Constitutional, other (General disorders) | 2 (5) | 1 (1) | 3 (3) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (34) | 11 (27) | 11 (23) | 12 (22)
creatinine (Hepatobiliary disorders) | 1 (4) | 5 (8) | 0 (0) | 8 (21)
Depression (Psychiatric disorders) | 3 (18) | 4 (15) | 3 (12) | 13 (28)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 12 (31) | 12 (30) | 20 (58) | 14 (32)
Dizziness (Nervous system disorders) | 6 (7) | 5 (6) | 3 (6) | 5 (5)
Dry Eye Syndrome (Eye disorders) | 0 (0) | 1 (8) | 2 (9) | 2 (5)
Dry Mouth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (11)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 4 (10) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (28) | 7 (26) | 8 (33) | 5 (11)
Dyspepsia (Gastrointestinal disorders) | 9 (28) | 5 (16) | 3 (17) | 7 (30)
Edema limb (Blood and lymphatic system disorders) | 5 (15) | 7 (29) | 5 (17) | 5 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1) | 0 (0) | 3 (5)
Extrapyramidal movement (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 14 (43) | 9 (53) | 8 (34) | 6 (18)
fatigue (General disorders) | 21 (117) | 29 (147) | 29 (149) | 29 (182)
febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
fever w/o neutropenia (General disorders) | 5 (6) | 7 (13) | 3 (3) | 4 (4)
flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (5)
Gastrointestinal-other (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (7) | 3 (5)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 37 (170) | 38 (191)
Head/headache (Nervous system disorders) | 31 (121) | 28 (99) | 23 (106) | 26 (113)
hematologic-other (Blood and lymphatic system disorders) | 3 (13) | 9 (108) | 4 (14) | 10 (51)
hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 9 (58) | 3 (8) | 5 (12)
hemorrhage-other (Blood and lymphatic system disorders) | 2 (7) | 2 (2) | 0 (0) | 2 (2)
hemorrhoids (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (4) | 0 (0)
Hot flashes (General disorders) | 16 (89) | 10 (78) | 11 (58) | 18 (72)
hypercalcemia (Metabolism and nutrition disorders) | 3 (13) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 12 (28) | 9 (23) | 7 (12) | 10 (39)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (5) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (9) | 4 (5) | 2 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (7) | 1 (4) | 4 (24) | 2 (6)
Hypertension (Blood and lymphatic system disorders) | 22 (50) | 16 (66) | 14 (54) | 14 (44)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (17) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (14) | 4 (5) | 1 (1) | 5 (6)
Hypoglycemia (Endocrine disorders) | 3 (3) | 4 (6) | 2 (2) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 6 (14) | 1 (1) | 0 (0) | 2 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (11) | 6 (10) | 0 (0) | 2 (10)
Infection Gr0-2 neut, bronchus (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Infection Gr0-2 neut, sinus (Infections and infestations) | 4 (7) | 3 (3) | 5 (10) | 3 (4)
Infection Gr0-2 neut, skin (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 2 (2)
Infection Gr0-2 neut, upper airway (Infections and infestations) | 5 (5) | 3 (4) | 6 (11) | 1 (1)
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 2 (3) | 1 (2) | 2 (4) | 1 (1)
Infection w/unk ANC upper airway NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Infection-other (Infections and infestations) | 8 (9) | 4 (4) | 1 (2) | 4 (6)
Insomnia (General disorders) | 8 (48) | 6 (19) | 9 (45) | 10 (44)
irregular menses (Reproductive system and breast disorders) | 2 (8) | 0 (0) | 1 (5) | 2 (3)
joint, pain (Musculoskeletal and connective tissue disorders) | 31 (156) | 18 (110) | 23 (111) | 24 (103)
joint-function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (5)
Leukocytes (Blood and lymphatic system disorders) | 9 (23) | 11 (34) | 4 (6) | 7 (19)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 2 (3)
Metabolic/laboratory-other (Metabolism and nutrition disorders) | 12 (42) | 12 (67) | 4 (7) | 5 (11)
Muco/stomatitis(symptom) oral cavity (Infections and infestations) | 9 (29) | 10 (43) | 20 (56) | 14 (36)
Muco/stomatitis by exam, oral cavity (Infections and infestations) | 1 (1) | 5 (22) | 8 (13) | 7 (9)
Muscle, pain (Musculoskeletal and connective tissue disorders) | 10 (28) | 4 (11) | 6 (13) | 4 (20)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (29) | 6 (16) | 5 (8)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (12) | 1 (2) | 2 (8)
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 5 (23)
Nausea (Gastrointestinal disorders) | 10 (23) | 19 (37) | 13 (27) | 17 (41)
Neck,pain (Musculoskeletal and connective tissue disorders) | 8 (14) | 1 (1) | 3 (4) | 4 (8)
Neuropathy-sensory (Nervous system disorders) | 10 (48) | 11 (47) | 11 (45) | 15 (58)
Neutrophils (Blood and lymphatic system disorders) | 6 (12) | 13 (26) | 4 (4) | 7 (17)
Nonneuropathic generalized weakness (General disorders) | 2 (11) | 0 (0) | 0 (0) | 1 (1)
Nose, hemorrhage (Blood and lymphatic system disorders) | 16 (45) | 19 (54) | 12 (28) | 14 (40)
Oral cavity, hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (3) | 3 (4)
Oral gums, pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pain NOS (Nervous system disorders) | 2 (9) | 0 (0) | 0 (0) | 0 (0)
Pain-other (Nervous system disorders) | 6 (15) | 9 (16) | 6 (12) | 7 (10)
Palpitations (Cardiac disorders) | 2 (5) | 2 (7) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 2 (9) | 4 (14) | 4 (8) | 5 (22)
Proteinuria (Renal and urinary disorders) | 21 (61) | 28 (89) | 25 (77) | 21 (71)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 (8) | 2 (3) | 2 (5) | 5 (7)
Pulmonary/upper respiratory-other (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 12 (43) | 10 (26) | 16 (44)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (12) | 8 (12) | 5 (9) | 3 (5)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (5) | 8 (12)
Rectum, hemorrhage (Gastrointestinal disorders) | 4 (9) | 0 (0) | 1 (1) | 0 (0)
Rigors/chills (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 2 (3) | 0 (0)
Skin-other (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 6 (12) | 7 (13)
Sweating (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (12) | 0 (0) | 1 (1)
Taste disturbance (General disorders) | 7 (27) | 4 (15) | 7 (36) | 8 (29)
Tearing (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Throat/Pharynx/larynx,pain (General disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Vagina, hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (4)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 2 (3) | 2 (3) | 1 (2) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 6 (19) | 1 (1) | 1 (1) | 2 (2)
Vision-blurred (Eye disorders) | 1 (1) | 2 (3) | 3 (5) | 1 (1)
Voice changes/dysarthria (General disorders) | 4 (14) | 5 (36) | 3 (8) | 2 (13)
Vomiting (Gastrointestinal disorders) | 7 (12) | 3 (6) | 6 (7) | 9 (13)
Weight Gain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (6)
Wound-non-infectious (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cardiac-other (Cardiac disorders) | 1 (3) | 3 (7) | 3 (4) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No